CLINICAL TRIAL: NCT02671747
Title: Pilot Testing for Mind Over Matter: Healthy Bowels, Healthy Bladder
Brief Title: Pilot: Mind Over Matter: Healthy Bowels, Healthy Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-0942
Record Dates: First submitted 2016-01-29; First posted 2016-02-02 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Urinary Incontinence; Fecal Incontinence; Accidental Bowel Leakage
MeSH Terms: conditions — Urinary Incontinence; Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pilot workshop (Experimental): Participants attend intervention. No control arm
  Interventions: Behavioral: Mind Over Matter; Healthy Bowels, Healthy Bladder

INTERVENTIONS:
Behavioral: Mind Over Matter; Healthy Bowels, Healthy Bladder — 3 workshop sessions over a one-month period using self-efficacy and health behavior change to improve incontinence symptoms and promote care-seeking if symptoms do not improve sufficiently

SUMMARY:
The study is to pilot-test an innovative, combined urinary/bowel continence workshop in two Wisconsin communities. Between 8-15 women with incontinence will be enrolled in each of the two pilot communities and will complete three 90-minute workshop sessions over a 6 week period.

DETAILED DESCRIPTION:
The pilot study will use mixed methods to compare pre- and post-workshop data about urinary and bowel incontinence symptoms and care-seeking from workshop participants as well as information about workshop acceptability from workshop participants and community partners. The study is expected to last 6 months from initial IRB approval through data analysis and workshop revision. This research will provide preliminary data for a larger test of this workshop in four diverse Wisconsin Communities, followed by a randomized, controlled trial and subsequent dissemination research study.

ELIGIBILITY:
Inclusion Criteria:

* qualifying symptoms in 3 months prior to enrollment

Exclusion Criteria:

* receiving new treatment for qualifying symptoms in 3 months prior to enrollment

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
urinary incontinence symptoms for participant with bladder symptoms | 3 months after workshop completion
  1. Change in Urinary Distress Inventory-6 Subscale of Pelvic Floor Distress Inventory-20 from baseline
  2. Patient Global Impression of Improvement in urinary symptoms at 3 month follow up
bowel incontinence symptoms for participant with bowel symptoms | 3 months after workshop completion
  1. Change in Colorectal Anal Distress Inventory-8 Subscale of Pelvic Floor Distress Inventory-20 from baseline
  2. Patient Global Impression of Improvement in bowel symptoms at 3 month follow up

SECONDARY OUTCOMES:
geriatric self-efficacy score for urinary incontinence | 3 months after workshop completion
  Difference between baseline and 3 month follow up on Geriatric Self-Efficacy for Urinary Incontinence scale
barriers to care-seeking for urinary incontinence | 3 months after workshop completion
  Score on the Barriers to Incontinence Care-Seeking Questionnaire (BICS-Q) at three month follow up as compared to baseline
barriers to care-seeking for accidental bowel leakage | 3 months after workshop completion
  Barriers to Care-Seeking for Accidental Bowel Leakage responses - difference from baseline to 3 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Brown, MD, Principal Investigator — University of Wisconsin, Madison

IPD SHARING:
Plan to Share IPD: Yes